## INFORMED CONSENT FORM COVER PAGE

## Study Title:

Effects of a Physical Activity Program for Children with Autism on Psychomotor and Psychosocial Characteristics

Principal Investigator: Ebru AYAZ

Independent Researcher / Kocaeli – Turkey

E-mail: ebrukaracar41@hotmail.com

Orcid: https://orcid.org/0009-0006-7186-9178

Second Author: Dilara Fatoş ÖZER

Istanbul Bilgi University / Faculty of Health Sciences - Department of Child Development /

Istanbul – Turkey

E-mail: dilara.ozer@bilgi.edu.tr

Orcid: https://orcid.org/0000-0001-5753-3332

Third Author: Gülsüm HATİPOĞLU ÖZCAN

Istanbul University-Cerrahpaşa / Faculty of Sport Sciences / Istanbul – Turkey

E-mail: gulsumhatipoglu@hotmail.com

Orcid: https://orcid.org/0000-0003-1059-8424

NCT Number: Not Yet Appointed

Document Type: Informed Consent Form

Document Date: 03/04/2022

## INFORMED CONSENT FORM

Information About the Study:

Study Title: Effects of a Physical Activity Program for Children with Autism on Psychomotor and Psychosocial Characteristics

Study Content: This study will include a total of 40 children diagnosed with autism spectrum disorder, consisting of 20 experimental and 20 control groups, aged 8-12, who are educated in special education application schools affiliated with the Kocaeli Provincial Directorate of National Education. The impact of the Physical Activity Program on the motor skills, psychosocial characteristics, quality of life, and physical fitness of children with autism will be examined. The impact of the Physical Activity Program on the motor skills, psychosocial characteristics, quality of life, and physical fitness of children with autism will be examined.

Research Objective: This study aims to examine the effects of the Physical Activity Program on the motor skills, social skills, and quality of life of children diagnosed with ASD. This approach will examine the physical activity levels of individuals with autism and develop recommendations on the necessary conditions for activity and the situations in which these conditions can be met.

Nature of the Research: This study will use a mixed-method sequential exploratory design consisting of two phases: quantitative and qualitative. The purpose of this design, which favors two patterns in a single study, is to ensure a more detailed and comprehensive understanding of a phenomenon by utilizing the advantages of both qualitative and quantitative patterns. In the quantitative phase, which evaluates the effect of the physical activity program (PAP) on psychomotor and psychosocial characteristics, an unequal pre-test-post-test control group design, which is part of the quasi-experimental model of quantitative research methods, will be used.

Expected Duration of the Study: Total duration 6 months.

Expected Number of Participants in the Study: 40

Procedures to be Followed in the Research: Within the scope of the research, the Gilliam Autism Spectrum Disorder Rating Scale-2-TV (GASDRS-2-TV), Quality of Life Scale (QOLS), Bruininks Oseretsky Motor Proficiency Test, Eurofit Test Battery, and Social Skills Rating System will be used for the experimental group and control group within the scope of the research. Test data will be entered at the beginning and end of the research, and the pre-test and post-test results of the two groups will be compared at the end of the application process. Face-to-face meetings with students are listed for planning group interviews focusing on qualified research methods regarding the physical activity level of the autistic child. During the interview, factors affecting the participation of children with autism spectrum disorder in physical activities will be discussed Ten questions explaining parental views will be answered. Interviews will be conducted after the consent form is signed. Each interview will last 60-90 minutes.

Voluntary Participation, Right to Refuse or Withdraw from the Study, Withdrawal from the Study:

- a. I give my permission for my child to participate in the study voluntarily, without any pressure or coercion.
- b. I have been informed that my child has the right to refuse to participate in the study at any time during the research process.
- c. I have been informed that my child may withdraw from the study at any time without giving any reason and without suffering any harm as a result of withdrawing from the study, provided that the responsible researcher is notified.

Confidentiality: The results of the study may be presented at scientific meetings or in publications. However, in such cases, your child's identity will be kept strictly confidential.

Consent to Participate in the Study: I have read the text titled "Informed Consent Form" above/had it read to me. The content and meaning of this information have been explained to me. I was given the opportunity to ask all the questions that came to mind and received satisfactory answers to my questions. Under these conditions, I agree to my child's voluntary participation in the study without any pressure or coercion.

I have received a signed copy of this document.

Signature: Mission:

Date:

| Parent's Name and Surname: | Researcher's Name and Surname: |
|----------------------------|--------------------------------|
| Age and Gender: | Signature: |
| Signature: | Date: |
| Address: | |
| Phone: | |
| Email: | |
| Date: | |
| Name and Surname: | |